CLINICAL TRIAL: NCT03136523
Title: Evaluation of the Prognostic and Predictive Significance of EGFR, Kirsten Rat Sarcoma (KRAS), Anaplastic Lymphoma Kinase , Programmed Death-Ligand 1 (PD-L1) Protein and Microsatellite Instability (MSI) in Lung Cancer
Brief Title: Tissue Microarrays (TMAs) Construction in Lung Cancer Samples
Acronym: LUNGTMA
Status: Completed | Type: Observational
Sponsor: Kostas N.Syrigos (Other)
Responsible Party: Sponsor-Investigator, Kostas N.Syrigos, PROFESSOR, Oncology Center of Biochemical Education And Research
Organization: Oncology Center of Biochemical Education And Research (Other)
Other Study IDs: D5162C00012; ESR-15-11047 (Other Grant/Funding Number: Astrazeneca S.A.)
Record Dates: First submitted 2017-04-21; First posted 2017-05-02 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Lung Cancer
Keywords: NSCLC; SCLC; MOLECULAR BIOMARKERS; EGFR; PD-L1; ALK; KRAS
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue samples from small biopsies ( core needle biopsy, FNB, excisional biopsy, incisional biopsy) or surgical resection
Oversight: Data Monitoring Committee: No

SUMMARY:
Construction of a large cohort of lung cancer patients to evaluate the Prognostic and Predictive Significance of the molecular biomarkers Epidermal growth factor receptor (EGFR), KRAS, Anaplastic lymphoma kinase (EML4-ALK), Programmed Death-Ligand 1 (PD-L1) protein and Microsatellite Instability (MSI) in lung cancer: A tissue microarray-based study of 500 cases.

DETAILED DESCRIPTION:
Research hypothesis The research hypothesis for this study is that the expression/status of various molecular biomarkers (mainly including EGFR, KRAS, ALK, PD-L1 and MSI) may confer additional prognostic ( in terms of disease outcome i.e. PFS and OS) and/or predictive ( in terms of treatment response) information for lung cancer patients.

The research hypothesis is reflected in the primary objective of this study, which is to further evaluate the prognostic and predictive significance of currently existing molecular markers (EGFR, KRAS, ALK, PD-L1 and MSI), as well as of future biomarkers that may evolve. Secondary objectives include the evaluation of the differential expression/status of the examined biomarkers (EGFR, KRAS, ALK, PD-L1 and MSI) and standard clinicopathologic parameters including: PFS, OS and treatment response as well as age, gender, smoking history/status, performance status (PS), serum lactate dehydrogenase (LDH) and albumin levels, disease stage, tumor size, histology and grade, presence or absence of brain metastases, presence or absence of liver metastases and number of metastatic sites (all at diagnosis), and treatment data (type of treatment(s) received and treatment response. Potential correlations/interactions between the examined biomarkers will also be explored.

Rationale for conducting this study Rationale for biomarker selection The primary aim of this study is to further clarify the differential expression/status and frequency of EGFR and KRAS mutations, ALK rearrangements, PD-L1 protein and MSI, as well as their association with various clinicopathologic parameters, including treatment response, progression-free survival (PFS) and overall survival (OS), in a large and heterogeneous cohort of patients with lung cancer (including both NSCLC and SCLC).

EGFR, KRAS and ALK are among the most clinically important biomarkers of treatment response in NSCLC; EGFR and ALK represent major therapeutic targets in NSCLC. However, relatively little is known as regards their expression and potential clinical significance in SCLC.

PD-L1 protein represents a candidate biomarker of prognosis as well as therapeutic target. Previous experimental and clinical research data have strongly suggested that immune check point inhibitors, including anti-PD-1 and anti-PD-L1 agents, may increase tumor cell vulnerability to immune destruction and potentially improve survival of patients with lung cancer. The MSI phenotype may also affect prognosis of NSCLC patients and response to treatment, including immune checkpoint blockade with PD-1 inhibitors.

Rationale for the use of TMAs TMA-based immunohistochemistry represents an innovative diagnostic approach with several important advantages as compared to conventional immunohistochemical methods. As widely acknowledged, the main and foremost advantage of this technology is its impressive potential to maximize and preserve tissue resources. Moreover, it provides an efficient and cost-effective alternative to conventional histopathologic processing for the performance of large-scale analyses with considerable savings in time, labor, reagents and other laboratory consumables [31]. Most importantly, and aside from cost reductions alone, another advantage of the TMA technique is the identical treatment of all studied samples. Since TMAs contain multiple tissue samples on a single slide, all these specimens are simultaneously subjected to the exact same environmental and experimental conditions (i.e. temperature, reagents concentration, incubation time, antigen retrieval procedure). This stands in sharp contrast to the substantial slide-to-slide variability associated with individual processing of whole tissue sections, thus underlying the superior standardization of the TMA technology [30].

Briefly, construction of TMAs will allow for simultaneous analysis of a large number of biomarkers, either at the protein or at the RNA level.

Benefit/risk and ethical assessment Potential risks and benefits As this is a non-interventional study, there are no physical potential risks to participants, other than potential breach of confidentiality; for the same reason, there are no potential benefits to participants.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Age >18 years at study enrollment
3. Histologically confirmed NSCLC or SCLC
4. Availability of and access to patients' medical records containing demographic, clinical and treatment data as of lung cancer diagnosis and until the date of patient registration in the study.
5. Representative formalin-fixed paraffin-embedded tissue blocks.

Exclusion Criteria:

1. Significant life-limiting comorbidity (such as end-stage cardiac, renal, pulmonary or liver disease)
2. Second concomitant malignancy or prior history of other malignancies
3. Known immunodeficiency .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be performed in a tertiary hospital and will include a cohort of patients, alive or deceased at the time of their registration in this study, with consecutive lung cancer diagnosis (adeno- and nonadeno- NSCLC and SCLC) between January 1, 2012 and December 31, 2015. A total number of 500 cases will be studied. The planned number of cases to be included in this translational study, has been estimated on the basis of the average actual number of lung cancer diagnoses handled by the Institutional pathological laboratory annually. The study populations will include 200 patients with lung adenocarcinoma, 150 patients with NSCLC (other than adenocarcinoma) and 150 patients with SCLC.
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
A translational research study of exploratory and descriptive nature of biomarkers in patients with lung cancer | The study is expected to start in the first quarter of 2016 and to end by the second quarter of 2019.
  500 cases will be studied. Three TMAs in total of lung adenocarcinoma, non-adenocarcinoma and SCLC, respectively- will be constructed. IHC for PD-L1 will be performed using commercially available antibodies and automated procedure. The EGFR, KRAS, ALK and MSI status will be assessed using routine molecular assays and procedures, either on the original FFPE tissue blocks or the constructed TMAs. MSI status will be evaluated using PCR-based method in FFPE tissue blocks. If that is not possible the status will be evaluate using IHC for the mismatch repair genes (MMR) hMLH1 and hMSH2 proteins expression on the TMAs. Biomarker characterization will be done according to the method that it will be used. For PD-L1: positive versus negative, for EGFR: mutant versus wild-type, for KRAS: mutant versus wild-type, for ALK: positive for ALK rearrangement versus negative for ALK rearrangement and for MSI: MSI high, MSI low, MSI stable.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos N Syrigos, MD,PhD, Principal Investigator — Non-Governmental, Non-Profit Organization
Locations (1):
- OCEBER, Athens, Greece

IPD SHARING:
Plan to Share IPD: No